CLINICAL TRIAL: NCT00274053
Title: Effect of a 9-month Treatment of SPIRIVA® on Health Related Quality of Life in Patients With Chronic Obstructive Pulmonary Disease. Validation of a New HRQoL Questionnaire Appropriate to Common Daily Practice. (TIPHON Study)
Brief Title: Effects of a 9-months Treatment of SPIRIVA on Health Related Quality of Life in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.256
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: tiotropium

SUMMARY:
The purpose of this study is to investigate the effect of a 9-month treatment of tiotropium (SPIRIVA®) 18 mcg once daily on Health Related Quality of Life and lung function in patients with a Chronic Obstructive Pulmonary Disease.

DETAILED DESCRIPTION:
This was a multicentre, randomised, double blind, parallel group, placebo-controlled, 9 month study. It was designed to determine the effect of inhaled tiotropium treatment on quality of life in patients with COPD.

Following an initial 2-week screening period, patients were randomized to either tiotropium or placebo at Visit 2. Patients returned to the clinic at month 3 (Visit 3), 6 (Visit 4), and 9 (Visit 5) for the conclusion of the trial. The patients received treatment daily for 9 months.

Quality of life was measured on each visit by using the Saint george's respiratory Questionnaire. Additionally a short form questionnaire was developped for that study (Visual Simplified Respiratory Questionnaire). Lung function was also measured at each visit by spirometry.

Study Hypothesis:

The primary objective of this study is to compare the efficacy of Tiotropium and placebo on improving HRQoL evaluated by the percentage of SGRQ responders. The null hypothesis is that there is no difference in the effect on HRQoL assessed by the percentage of SGRQ responders between the two treatment groups. The alternative hypothesis is that there is a difference in effect on HRQoL assessed by the percentage of SGRQ responders between tiotropium and placebo. The test will be performed at the alpha = 0.05 level of significance.

Comparison(s):

Tiotropium 18 mcg once daily vs Placebo

ELIGIBILITY:
Diagnosis of COPD and matching the following criteria:

* Baseline 20 % < FEV1 < 70 % of European Community of Coal and Steel (ECCS) predicted values .
* Baseline FEV1/SVC< 70 %. Smoking history > 10 pack-years (p.y.). A p.y. was defined as the equivalent of smoking one pack of cigarettes per day for one year.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2002-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04

PRIMARY OUTCOMES:
responder rate on SGRQ questionnaire (% of patients improved by more than 4 points)

SECONDARY OUTCOMES:
changes in SGRQ scores, VSRQ scores, spirometric parameters (FEV1, FVC, FIV1, SVC, IC) ; incidence, severity and duration of acute exacerbations, PGE

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BI France S.A.S.
Locations (27):
- France (27):
  - Boehringer Ingelheim Investigational Site, Aix-les-Bains
  - Hôpital Privé Antony, Antony
  - Boehringer Ingelheim Investigational Site, Bordeaux
  - Boehringer Ingelheim Investigational Site, Cambo-les-Bains
  - Centre Médical Annie Enia, Cambo-les-Bains
  - Boehringer Ingelheim Investigational Site, Châlons Sur Saône
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Boehringer Ingelheim Investigational Site, Colmar
  - CH Laennec, Creil
  - Boehringer Ingelheim Investigational Site, Dole
  - Centre Hospitalier, Longjumeau
  - Boehringer Ingelheim Investigational Site, Lunéville
  - MAPI CRO, Lyon
  - Boehringer Ingelheim Investigational Site, Maxéville
  - Boehringer Ingelheim Investigational Site, Metz
  - Hôpital Notre Dame de Bon Secours, Metz
  - Boehringer Ingelheim Investigational Site, Montigny-lès-Metz
  - Boehringer Ingelheim Investigational Site, Mulhouse
  - Hôpital Pitié Salpétrière, Paris
  - Hôpital Cochin, Paris
  - Boehringer Ingelheim Investigational Site, Poitiers
  - Hôpital Saint Charles, Saint-Dié
  - Groupe Hospitalier Sud Réunion, Saint-Pierre
  - Boehringer Ingelheim Investigational Site, Saint-Quentin
  - CH Toul, Toul
  - Boehringer Ingelheim Investigational Site, Toulouse
  - Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy